CLINICAL TRIAL: NCT02619513
Title: Effects of Dexmedetomidine as an Adjunctive Analgesic Used in Continuous Thoracic Paravertebral Blocks for Post-thoracotomy Pain Syndrome
Brief Title: Effects of Dexmedetomidine Used in Continuous Thoracic Paravertebral Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weifeng Tu (Other)
Responsible Party: Sponsor-Investigator, Weifeng Tu, Chief Physician, Guangzhou General Hospital of Guangzhou Military Command
Organization: Guangzhou General Hospital of Guangzhou Military Command (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Dexmedetomidine TPVB
Record Dates: First submitted 2015-09-22; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Post-thoracotomy Pain Syndrome
Keywords: Paravertebral Blocks; Dexmedetomidine; Analgesia; Inflammatory response; Thoracotomy
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- General anesthesia group(Group GA) (No Intervention): Group GA received general anesthesia only and intravenous analgesia pump.
- TEB group(Group GE) (Experimental): Group GE received continuous thoracic epidural block(TEB) combined with general anesthesia and postoperative continuous thoracic epidural analgesia, and only added ropivacaine in PVB as an postoperative adjuvant.
  Interventions: Drug: Ropivacaine
- PVB without DEX group (Group GT) (Experimental): Group GT received ultrasound-guided(Mindray M7 series) continuous thoracic paravertebral nerve block(PVB) combined with general anesthesia and continuous thoracic paravertebral nerve block patient-controlled analgesia, and only added ropivacaine in PVB as an postoperative adjuvant.
  Interventions: Drug: Ropivacaine; Device: Mindray M7 series
- PVB with DEX group(Group GTD) (Experimental): Group GTD received ultrasound-guided(Mindray M7 series) continuous thoracic paravertebral nerve block combined with general anesthesia and continuous thoracic paravertebral nerve block patient-controlled analgesia,but with dexmedetomidine 0.5μg/kg added to ropivacaine in PVB as an adjuvant.
  Interventions: Drug: Dexmedetomidine; Drug: Ropivacaine; Device: Mindray M7 series

INTERVENTIONS:
Drug: Dexmedetomidine — Group GTD received thoracic continuous paravertebral nerve block with dexmedetomidine (0.5μg/kg) added to ropivacaine before anesthesia induction, and used continuous thoracic paravertebral nerve block patient-controlled analgesia(with dexmedetomidine 100μg）.
  Arms: PVB with DEX group(Group GTD)
Drug: Ropivacaine — Group GE\GT\GTD respectively received continuous nerve blocks and postoperative analgesia combined with ropivacaine.
  Arms: PVB with DEX group(Group GTD); PVB without DEX group (Group GT); TEB group(Group GE)
Device: Mindray M7 series — Ultrasound real-time guidance have been used in continuous thoracic paravertebral blocks in group GT and group GTD.
  Arms: PVB with DEX group(Group GTD); PVB without DEX group (Group GT)

SUMMARY:
The purpose of this study is to explore the effectiveness of dexmedetomidine as an adjunctive analgesic, used in ultrasound-guided continuous thoracic paravertebral blocks for Post-thoracotomy Pain Syndrome(PTPS).

DETAILED DESCRIPTION:
Thoracic surgical procedures are among the most painful operations, and their outcomes are affected adversely by postoperative discomfort. Post-thoracotomy pain syndrome (PTPS) is a well-recognized complication of thoracotomy. Post-thoracotomy pain control improves patient satisfaction and decreases postoperative complication morbidity. Epidural analgesia used to be considered as the best method of pain relief after major surgery despite its side-effects, which includes hypotension, respiratory depression, incomplete or failed block, etc. Recently, paravertebral block is an alternative technique that may offer a comparable analgesic effect and a better side-effect profile for post-thoracotomy pain. Dexmedetomidine(DEX) is a Food and Drug Administration-approved, parenteral, selective α2-agonist that induces anxiolytic and analgesia without respiratory depression. It could provide dose-dependent sedation , analgesia , anti-anxiety and inhibition of sympathetic nerves and other effects . Current studies with regard to the effectiveness of DEX as an adjunctive medicine, used in ultrasound-guided continuous thoracic paravertebral blocks for PTPS. The mechanical withdrawal threshold and VAS scores are recorded. The consumption of opioid and general anesthetics during perioperative period are also recorded. To compare the incidence rates of side effects, such as nausea, vomiting, dizziness, hypotension and bradyarrhythmia in the first 3 days after operation among the groups.Also,to measure and compare the level of inflammatory factor in different group.A questionnaire is adopted to investigate whether there are chronic pain symptoms happen at 6 months after the operation which aim to PTPS.

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ⅰ～Ⅲ patient undergoing thoracotomy;
2. Written informed consent from the patient or the relatives of the participating patient.
3. BMI:18～25kg/m2

Exclusion Criteria:

1. Mental illness;
2. Epidural anesthesia or thoracic paravertebral blocks contraindicated;
3. People who have Slow-type arrhythmias or hypotension;
4. People who have lung infection or sleep apnea syndrome;
5. People who have chronic renal failure;
6. Alcohol or drug abuse;
7. Already taking gabapentin, pregabalin, benzodiazepin or antidepression drug;
8. Local anesthetics allergy;

Ages: 19 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Baseline mechanical withdrawal threshold(unit: g) of patients without treatment-related events. | the day before the operation
  Baseline quantization degree of algesia without treatment-related events before receiving thoracotomy measured by Electric Von Frey 2391, and the testing position is located in the intercostal skin at the level of operation incisions, which about 2cm away from the incision.
The change of mechanical withdrawal threshold(unit: g) of patients with different treatment-related events in the following one week after thoracotomy. | 12, 24, 48, 72h and 1w after the operation
  To show the changing trend of quantization degree of hyperalgesia and allodynia with different treatment-related events after receiving thoracotomy measured by Electric Von Frey 2391, and the testing position is located in the intercostal skin at the level of operation incisions, which about 2cm away from the incision.
The change of Interleukin-6(IL-6) of patients with different treatment-related events during the perioperative period. | pre-operation and 6, 24, 72h after the operation
  The changing trend of plasma IL- 6 in venous blood of patients with different treatment-related events during the perioperative period. And the blood time is in the morning before patients feed at each expected testing time point.
The change of Interleukin-10(IL-10) of patients with different treatment-related events during the perioperative period. | pre-operation and 6, 24, 72h after the operation
  The changing trend of plasma IL-10 in venous blood of patients with different treatment-related events during the perioperative period. And the blood time is in the morning before patients feed at each expected testing time point.
The change of tumor necrosis factor-α(TNF-α) of patients with different treatment-related events during the perioperative period. | pre-operation and 6, 24, 72h after the operation
  The changing trend of TNF-α in venous blood of patients with different treatment-related events during the perioperative period. And the blood time is in the morning before patients feed at each expected testing time point.

SECONDARY OUTCOMES:
The change of visual analogue scale(VAS) of patients with different treatment-related events in the following one week after thoracotomy. | 12, 24, 48, 72h and 1w after the operation
  To show the changing trend of visual analogue scale(VAS) in order to subjectively speculate the degree of hyperalgesia and allodynia with different treatment-related events after receiving thoracotomy, and the testing position is located in the intercostal skin at the level of operation incisions, which about 2cm away from the incision.
The intraoperative consumption of opioids. | From the beginning to the end of the anesthesia procedure.
  The consumption of opioid(remifentanil and sufentanil) during the operation are recorded(the consumption of sufentanil was converted to the consumption of remifentanil producing the equivalent effect by 1:10,unit:mg).
The postoperative consumption of opioids. | in the first 3 days after operation
  If insufficient analgesia happens(resting VAS scores>4), than use dezocine intravenously as additional analgesia(a single dose 5-20mg, no more than 120mg per day). The consumption of opioid(dezocine) in the following 3 days after the operation are recorded(unit:mg).
The change of mean arterial pressure (MAP) of the patients when receiving the thoracotomy. | the key time have been distributed into five parts: when the patient was brought to the operation room (T0), 15 mins after paravertebral administration (T1), after intubation (T2), after skin incision (T3), before extubation (T4)
  To show the changing trend of hemodynamics with different treatment-related events when receiving thoracotomy.
The change of heart rate(HR) of the patients when receiving the thoracotomy. | the key time have been distributed into five parts: when the patient was brought to the operation room (T0), 15 mins after paravertebral administration (T1), after intubation (T2), after skin incision (T3), before extubation (T4)
  To show the changing trend of hemodynamics with different treatment-related events when receiving thoracotomy.
The incidence rates of side effects. | in the first 3 days after operation
  To compare the incidence rates of side effects, such as nausea, vomiting, dizziness, hypotension and bradyarrhythmia in the first 3 days after operation.
A questionnaire related to postoperation chronic for the patients who have receiving thoracotomy. | at 6 months after operation
  A questionnaire is adopted to investigate whether there are chronic pain symptoms happen at 6 months after the operation which aim to PTPS.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Peng, PhD, Principal Investigator — Guangzhou General Hospital of Guangzhou Military Command
Locations (1):
- Department of Anesthesiology，Guangzhou Military Region General Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Ding X, Jin S, Niu X, Ren H, Fu S, Li Q. A comparison of the analgesia efficacy and side effects of paravertebral compared with epidural blockade for thoracotomy: an updated meta-analysis. PLoS One. 2014 May 5;9(5):e96233. doi: 10.1371/journal.pone.0096233. eCollection 2014. PMID 24797238
- [Background] Komatsu T, Sowa T, Takahashi K, Fujinaga T. Paravertebral block as a promising analgesic modality for managing post-thoracotomy pain. Ann Thorac Cardiovasc Surg. 2014;20(2):113-6. doi: 10.5761/atcs.oa.12.01999. Epub 2013 Feb 28. PMID 23445804
- [Background] Kimura M, Saito S, Obata H. Dexmedetomidine decreases hyperalgesia in neuropathic pain by increasing acetylcholine in the spinal cord. Neurosci Lett. 2012 Oct 31;529(1):70-4. doi: 10.1016/j.neulet.2012.08.008. Epub 2012 Aug 16. PMID 22917606
- [Background] El-Morsy GZ, El-Deeb A, El-Desouky T, Elsharkawy AA, Elgamal MA. Can thoracic paravertebral block replace thoracic epidural block in pediatric cardiac surgery? A randomized blinded study. Ann Card Anaesth. 2012 Oct-Dec;15(4):259-63. doi: 10.4103/0971-9784.101848. PMID 23041682